CLINICAL TRIAL: NCT02382185
Title: Non Invasive Cardiac Output Monitoring to Guide Goal Directed Fluid Therapy in High Risk Patients Undergoing Urgent Surgical Repair of Proximal Femoral Fractures
Acronym: ClearNOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: YOR-A02333
Record Dates: First submitted 2015-02-02; First posted 2015-03-06 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Hip Fractures
Keywords: Cardiac output
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Experimental): No intervention apart from application of clearsight monitor. Prior to induction of anaesthesia the control group will have a Clearsight cardiac monitor probe placed on a suitable finger and baseline haemodynamic measurements will be taken. All fluid management and administration of vasopressor therapy will be at the discretion of the anaesthetist as per the current practice at the host institution. Data on stroke volume, heart rate, blood pressure, cardiac output, oxygen saturations, will be recorded at baseline and then every 5 minutes.
  Interventions: Device: Application of clearsight monitor
- Fluid optimisation (Experimental): Application of clearsight monitor, optimisation of blood pressure and fluid optimisation. A Clearsight cardiac probe is attached and after induction of anaesthesia stroke volume is optimised using 250ml boluses of Hartmann's solution. The SV measurement prior to the final fluid bolus will be the optimal SV. Mean arterial blood pressure will be maintained within 30% of baseline values using a phenylephrine infusion.Data on haemodynamics will be recorded at baseline and then every 5 minutes, as well as before and after a fluid bolus. Haemoglobin will be maintained at>10g/dL with blood transfusion as required.
  Interventions: Other: Fluid optimisation; Drug: Optimisation of blood pressure; Device: Application of clearsight monitor

INTERVENTIONS:
Other: Fluid optimisation — The intervention will consist of optimising stroke volume with 250ml of Hartmanns solution
  Arms: Fluid optimisation
Drug: Optimisation of blood pressure — Phenylephrine infusion will be used to target a mean arterial blood pressure to within 30% of baseline (preoperative) value
  Arms: Fluid optimisation
Device: Application of clearsight monitor — The clear sight monitor will be applied to measure stroke volume.

SUMMARY:
Improving or maximising cardiac output in the perioperative setting through the use of goal directed fluid therapy has been shown to reduce complications and length of hospital stay in patients undergoing major abdominal surgery. The evidence for patients having surgery to repair a fractured neck of femur is less robust but many of these latter patients are elderly and often at high risk of complications.

Patients undergoing surgery (including surgery for hip fracture) under spinal anaesthesia have not had access to goal directed fluid therapy because of the invasive nature of the existing monitoring technology such as oesophageal doppler. The availability of a non invasive cardiac monitoring device, the Clearsight™, now makes goal directed fluid therapy a possibility for this group of patients.

This is a randomised controlled, observer blinded trial to assess the effects of goal directed fluid therapy in high-risk patients undergoing surgical repair of proximal femoral fractures.

The aim of the trial is to test the hypothesis that maximising circulating volume intra-operatively with balanced crystalloid reduces post-operative morbidity in high-risk patients undergoing urgent surgical repair of proximal femoral fractures.

DETAILED DESCRIPTION:
The management of fractured neck of femur in the elderly population is of clinical and political interest in the United Kingdom at present, with a current national audit in progress to look at anaesthetic management and clinical outcomes. It is estimated that the number of patients that sustain a hip fracture will reach 100,000 cases per annum by 2033 with a cost to the NHS of some £ 2.7 billion. Outcomes for this group remain poor with a mortality of 8% at 1 month, increasing to 20-33% at 1 year4. Complication rates for this group also remain significant with between 20 and 60% of patients having significant postoperative complications. These complications are not only associated with increased length of stay and healthcare costs, but also reduced long-term survival.

Improving or maximising cardiac output in the perioperative setting either through the use of intravenous fluids, or in combination with inotropes has been shown to reduce complication rates following surgery in a variety of settings including those with fractured neck of femurs. A recent meta analysis of optimisation trials has shown that for every 100 patients in whom the intervention is provided, patients will avoid a complication, and length of stay will be reduced by 1 day. Importantly the intervention is also associated with no harm. In 1997 by using the oesophageal Doppler to guide fluid therapy in an attempt to maximise cardiac output, Sinclair managed to reduce the time patients who were operated on for a fractured neck of femur were deemed fit for medical discharge from 15 to 10 days (P<0.05). Stroke volume was significantly increased in the protocol group, and although postoperative complication rates were not reported in this trial, it is inferred that they were reduced. A similar trial comparing conventional fluid therapy versus therapy guided by either central venous pressure measurements or oesophageal Doppler showed a similar reduction in time to being medically fit for discharge. This trial did report morbidity, which showed a non-significant trend to improvement in subjects who received oesophageal Doppler monitoring.

One of the main limitations of these trials are the relatively small numbers, with just 20 per group in the Sinclair trial and 30 per groups in the Venn trials, yet even with small numbers an improvement in outcome was seen. A larger trial has recently been completed using a more invasive calibrated measure of cardiac output, targeting a somewhat aggressive oxygen delivery of > 600ml/min/m2 using inotropic support in elderly fractured neck of femur patients. Few patients actually achieved this goal, however there was again a non-significant reduction in complications (RR 0.79, 95% CI 0.54-1.16) however the trial was underpowered due to issues with recruitment. The trial recruited 149 patients in total and to date is the largest study to examine this population despite the impact that this population has on the health services both within the NHS and worldwide. In addition all of the trials described included in their recruitment a broad group of patients some of whom could be considered to be at low risk of post operative complications.

Within this group of elderly patients a high-risk group exist. The Nottingham hip fracture score (NHFS) is a validated scoring system that predicts patients at increased risk of both 30 day and 1-year mortality. A NHFS ≥ 5 was associated with a mortality of 13.7% vs. 3.5% at 30 days (P<0.001) and 45.5% vs. 15.9% at 1 year (P<0.001). It is assumed that this high-risk group with an increased mortality rate also have an increased complication rate, and hence any effective intervention would have a greater impact on outcomes.

An increasing number of operations to repair fractured necks of femur are being performed awake under spinal anaesthesia. Technology such as oesophageal Doppler is not suitable as it cannot easily be tolerated when awake, and arterial based pulse waveform analysis requires an invasive procedure to be performed. Hence many patients do not receive goal directed therapy even though it may be of clinical benefit. A recent economic analysis has also suggested that goal directed therapy in this group is not only cost effective but also associated with cost savings.

The Clearsight™ non invasive cardiac output device measures blood pressure using the volume clamp method developed by the Czech physiologist Jan Penaz. Using a simple non-invasive finger cuff, the volume of an artery is kept clamped at a constant diameter. Changes in diameter are measured by a photo-plethysmograph within the finger cuff, and a servo controller applies counter pressure to keep the diameter of the artery constant. This allows the measurement of beat to beat blood pressure and hence cardiac output can also be calculated. The simple and non invasive nature of this device makes it suitable to use in patients undergoing repair of fractured neck of femur regardless of the type of anaesthetic. It requires no calibration, and would make goal directed therapy accessible to this group. The Clearsight has been shown to be a valid measure of cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* Patients due to undergo urgent or emergency repair of a proximal femoral fracture who have a Nottingham hip fracture score (NHFS) ≥ 5 i.e. patients who are regarded as 'high risk'.

Exclusion Criteria:

* Age < 50 years. Patients scoring 5 on the American Society of Anesthesiologists (ASA) physical status classification Multiple injuries requiring operative management

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Composite basket of complication | In hospital participants are expected to have a median hospital length of stay of 18 days
  The number of patients who develop one or more in hospital post operative complications as defined by Copeland (POSSUM) and modified for this patient group

SECONDARY OUTCOMES:
Incidence of major and minor complications | in hospital -Participants are expected to have a median hospital length of stay of 18 days
  Incidence of major and minor complications
Morbidity at day 3, 5, 10 measured by Post operative morbidity survey | 10 days
  Morbidity at day 3, 5, 10 measured by Post operative morbidity survey
Length of stay in hospital after surgery. | In hospital- participants are expected to have a median hospital length of stay of 18 days
  Length of stay in hospital after surgery.
time to drinking | in hospital - participants are expected to have a median hospital length of stay of 18 days
  time to drinking
time to eating | in hospital - participants are expected to have a median hospital length of stay of 18 days
  time to eating
time to mobilisation | in hospital - participants are expected to have a median hospital length of stay of 18 days
  time to mobilisation
Change ineri-operative haemodynamic variables - heart rate. | perioperative - from start of surgery to end
  Change ineri-operative haemodynamic variables - heart rate.
Change in peri-operative haemodynamic variables - blood pressure | perioperative - from start of surgery to end
  Change in peri-operative haemodynamic variables - blood pressure
Change in peri-operative haemodynamic variables - stroke volume | perioperative - from start of surgery to end
  Change in peri-operative haemodynamic variables - stroke volume
Incidence of perioperative hypotension. | perioperative
  Incidence of perioperative hypotension.
Total dose of administered vasopressor. | perioperative - from start of surgery to end
  Total dose of administered vasopressor.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Davies, MB FRCA MD, Principal Investigator — York Teaching Hospital
Locations (2):
- United Kingdom (2):
  - York Teaching Hospitals NHS Foundation Trust, York, North Yorkshire
  - Harrogate Hospital, Harrogate, Yorkshire

REFERENCES:
- [Derived] Davies SJ, Yates DR, Wilson RJT, Murphy Z, Gibson A, Allgar V, Collyer T. A randomised trial of non-invasive cardiac output monitoring to guide haemodynamic optimisation in high risk patients undergoing urgent surgical repair of proximal femoral fractures (ClearNOF trial NCT02382185). Perioper Med (Lond). 2019 Aug 8;8:8. doi: 10.1186/s13741-019-0119-x. eCollection 2019. PMID 31406569